CLINICAL TRIAL: NCT03208998
Title: The Changes of Natural Killer Cells Frequency and Function During Pegylated Interferon α-2a and Nucleoside Analogues Treatment in Patients With Chronic Hepatitis B.
Brief Title: The Changes of Natural Killer Cells Frequency and Function During Antiviral Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DTXY012
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis B Infection
Keywords: hepatitis B virus; Chronic Hepatitis B Infection; Pegylated Interferon α-2a; Nucleoside Analogues; Natural Killer Cells
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): patients who were untreated ever in immune-active phase were given subcutaneous injection of Peginterferon Alfa-2a with starting dose of 180 mg/weekly till 48 weeks.
  Interventions: Drug: Peginterferon Alfa-2a
- control group (No Intervention): patients who were untreated ever in immune-active phase took Nucleoside Analogues for maintenance treatment.

INTERVENTIONS:
Drug: Peginterferon Alfa-2a — patients untreated in immune-active phase were given subcutaneous injection of Peginterferon Alfa-2a with starting dose of 180 mg/weekly in experiment group.
  Other Names: Peg-IFN-α
  Arms: experimental group

SUMMARY:
Pegylated interferon α-2a(Peg-IFN-α) not only inhibit viral replication, but also play an important role in immune regulation, while Nucleoside analog(ue) drugs only inhibit viral replication. In hepatitis B infection, NKs are the main effector cells in early antiviral innate immune response. This study was aimed at investigating the changes of NKs frequency and function, and the expression of costimulatory molecules during Peg-IFN-αand nucleoside analog(ue) therapy.Meanwhile, investigators want to verify whether Peg IFN - alpha suppressed the virus and the reduction of virus led to the recovery of NKs function, or Peg IFN - alpha enhanced NKs function which gave rise to the decline of the virus.

DETAILED DESCRIPTION:
Pegylated interferon α-2a(Peg-IFN-α)and Nucleoside analog(ue) drugs can inhibit viral replication , but Peg-IFN-α also play an important role in immune regulation . In hepatitis B infection, NKs are the main effector cells in early antiviral innate immune response.Peg-IFN-α recommended as the first-line treatment has a higher chance to achieve HBeAg seroconversion and even HBsAg disappearance than nucleoside analog(ue) drugs, which may be related to the functional activation of pDCs in the case of hepatitis and the function enhancement of NKs during Peg-IFN-α therapy. This study was aimed at investigating the changes of NKs frequency and function, and the expression of costimulatory molecules during Peg-IFN-αand nucleoside analog(ue) therapy.Meanwhile, investigators want to explore whether the decline of HBsAg and HBeAg resulted in recovery of NKs function, or recovery of NKs function led to the decrease of HBsAg and HBeAg. Several studies demonstrated that HBsAg and HBeAg could damage NKs function, and the loss of HBsAg and HBeAg led to recovery of NKs function.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg and HBeAg positive for more than 6 months, HBV DNA detectable with ALT level abnormal lasted for three months and at least time190 IU/L or liver puncture biopsy demonstrated apparent inflammation, never treated before enrolled.

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the changes of Natural Killer Cells | at baseline and at treatment week 12, 24
  the changes of NK%,CD56bri/NK%,CD56dim/NK%,IFNAR2+NK%,IFNAR2MFI,NKp46+/NK%,NKp46dim/NK%,NKp46high/NK%, NKp46MFI,and NKp46ABC will be measured by flow cytometry during Pegylated Interferon α-2a and Nucleoside Analogues Treatment

SECONDARY OUTCOMES:
the change of HBVDNA levels (IU/ML) | at baseline and at treatment 12, 24, 36, 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBV markers and HBV DNA levels and liver function
the change of ALT levels(U/L) | at baseline and at treatment 12, 24, 36, 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBV markers and HBV DNA levels and liver function
the change of AST levels(U/L) | at baseline and at treatment 12, 24, 36, 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBV markers and HBV DNA levels and liver function

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Cao W, Li M, Zhang L, Lu Y, Wu S, Shen G, Chang M, Liu R, Gao Y, Hao H, Hu L, Yi W, Pan CQ, Xie Y. The Characteristics of Natural Killer Cells in Chronic Hepatitis B Patients Who Received PEGylated-Interferon versus Entecavir Therapy. Biomed Res Int. 2021 Jan 25;2021:2178143. doi: 10.1155/2021/2178143. eCollection 2021. PMID 33575322